CLINICAL TRIAL: NCT03002454
Title: A Cross-over Comparison of the Diagnostic Accuracy of Technetium (99mTc) Medronate Injection Prepared With 99mTc Derived From Neutron-activation Produced 99Mo Versus the Current Reference Standard of 99mTc Derived From Fission-produced 99Mo
Brief Title: Sodium Pertechnetate (99Tc) Injection Generator: 99mTc From Neutron-activation 99Mo v 99mTc From Fission 99Mo
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Altered biodistribution in investigational images versus standard images.
Sponsor: University of Manitoba (Other)
Collaborators: Winnipeg Regional Health Authority (Other)
Responsible Party: Principal Investigator, Dr. Sandor J. Demeter, Head, Nuclear Medicine, University of Manitoba
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NA 99Mo 001
Record Dates: First submitted 2016-12-12; First posted 2016-12-23 (Estimated); Results first posted 2017-10-03 (Actual); Last update posted 2017-10-03 (Actual); Status verified 2017-05

CONDITIONS: Cancer of Bone
Keywords: 99mTc Pertechnetate; Sodium Pertechnetate; Technetium; Molybdenum; MDP; neutron activation
MeSH Terms: conditions — Bone Neoplasms | interventions — Sodium Pertechnetate Tc 99m; Neutrons

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 99mTc MDP Injection:neutron-bombardment (Experimental): Oncologic indication for which a bone scan would normally be indicated. Participant having recently had a bone scan using Technetium (99mTc) Medronate Injection USP labeled with 99mTc derived from fission-sourced 99Mo. The images of the 99mTc MDP Injection-neutron-bombardment will be compared to the previous (on file) images from the 99mTc MDP Injection-fission
  Interventions: Drug: 99mTc MDP Injection:neutron-bombardment

INTERVENTIONS:
Drug: 99mTc MDP Injection:neutron-bombardment — Technetium (99mTc) Medronate Injection USP labeled with 99mTc derived from neutron-activation-produced 99Mo.
  Other Names: Sodium Pertechnetate (99Tc) Injection Generator (neutron)

SUMMARY:
A non-fission sourced, solvent generator produced 99mTc intravenous injection, as 99mTc -MDP, is to be used as a bone scan diagnostic radiopharmaceutical for assessment of bone pathology using the same oncologic indications as nuclear reactor sourced 99mTc, as 99mTc-MDP.

DETAILED DESCRIPTION:
This clinical trial will be a comparison of diagnostic and imaging equivalency of 99mTc Pertechnetate intravenous injection (labeled with commercial MDP kits) produced by a non-fission sourced/solvent generator and a nuclear reactor/column sourced generator. Each oncologic participant acts as their own control to reduce error variance.

Condition Intervention Phase Oncologic indication for which a bone scan would normally be indicated. Participant having recently had a bone scan using Technetium (99mTc) Medronate Injection USP labeled with 99mTc derived from fission-sourced 99Mo. Drug: Technetium (99mTc) Medronate Injection USP labeled with 99mTc derived from neutron-activation-produced 99Mo. Phase 3

ELIGIBILITY:
Inclusion Criteria:

* Oncology out-patients in whom an acceptable quality standard-of-care Technetium (99mTc) Medronate bone scan has been ordered or obtained within the last 28 days.
* If female of child-bearing potential is outside of the window of 10 days since the last menstrual period, a negative serum pregnancy test is required.
* Age greater than or equal to 18 years.

Exclusion Criteria:

* Oncology out-patients in whom an acceptable quality standard-of-care Technetium (99mTc) Medronate bone scan has been ordered or obtained within the last 28 days.
* If female of child-bearing potential is outside of the window of 10 days since the last menstrual period, a negative serum pregnancy test is required.
* Age greater than or equal to 18 years.
* Identified interval events which have occurred after the standard of care bone scan but prior to the administration of non-fission sourced Technetium (99mTc) Medronate which could influence or change bone scan uptake (e.g. skeletal trauma, orthopedic surgery, bone infection, or interval therapy (i.e. radiation therapy, non-maintenance chemotherapy). -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2016-08; Primary Completion 2016-11 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sandor J Demeter, MSc MD FRCPC, Principal Investigator — Winnipeg Regional Health Authority
Locations (1):
- Health Sciences Centre, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Oncologic bone imaging subjects screened and enrolled at Health Sciences Centre, Winnipeg, Manitoba from August to November 2017.
Pre-assignment Details: Previous bone imaging scan, within 3 to 28 days, using fission derived 99mTc MDP Injection to act as comparator for investigative drug (neutron-bombardment derived 99mTc MDP Injection) bone imaging scan of same subject.
Groups:
- 99mTc MDP Injection:Neutron-bombardment: Oncologic indication for which a bone scan would normally be indicated. All 4 participants initially had a bone scan using Technetium (99mTc) Medronate Injection USP labeled with 99mTc derived from fission-sourced 99Mo.
  3-28 days later all participants had a second bone scan using Technetium (99mTc) Medronate Injection USP labeled with 99mTc derived from neutron-activation-produced 99Mo.
Period: Overall Study
Arm/Group | 99mTc MDP Injection:Neutron-bombardment
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- 99mTc MDP Injection:Neutron-bombardment: Oncologic indication for which a bone scan would normally be indicated. Participant having recently had a bone scan using Technetium (99mTc) Medronate Injection USP labeled with 99mTc derived from fission-sourced 99Mo.
  99mTc MDP Injection:neutron-bombardment: Technetium (99mTc) Medronate Injection USP labeled with 99mTc derived from neutron-activation-produced 99Mo.
Arm/Group | 99mTc MDP Injection:Neutron-bombardment
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 1
Age, Continuous [Mean (Full Range); unit: years] | 61.5 [44 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 2
Region of Enrollment [Number; unit: participants]
  Canada | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Analyzed for Diagnostic Efficacy of Technetium (99mTc) Medronate Injection Prepared With 99mTc Derived From Neutron-activation Produced 99Mo Imaging Sensitivity Versus 99mTc Derived From Fission-produced 99Mo Imaging Sensitivity.
Description: All enrolled patients were re-imaged 3 to 28 days post a standard of care fission derived 99Mo bone scan using neutron-activation produced 99Mo as the investigational product. Per protocol dosage, time factors, injection site and imaging camera were matched. Resulting image sets (fission and neutron-activation) were analyzed visually for concordant biodistribution.
Time Frame: 60 days
Population: Each participant (4) acted as their own control to reduce variance. Paired image sets were analyzed visually for concordant biodistribution between the 99mTc Medronate Injection prepared with 99mTc derived from Neutron-activation produced 99Mo versus 99mTc Medronate Injection derived from Fission-produced 99Mo referenced as the baseline standard.
Measure: Count of Participants; unit: Participants
Arm/Group | 99mTc MDP Injection:Neutron-bombardment
Number analyzed (Participants) | 4
Participants | 4
Statistical Analysis 1: Comparison: 99mTc MDP Injection:Neutron-bombardment; Test type: Equivalence — Control: 99mTc MDP Injection:fission Investigation: 99mTc MDP Injection:neutron-bombardment Anticipated sample size of 50 participants with sample size parameters of: Alpha 0.05 Power 80% Kappa of significance 0.7 - 0.8 Prevalence of abnormal bone scans 30% Actual study population of 4 participants with 4 out of 4 demonstrating gross abnormal biodistribution therefore the study was terminated and no statistical analysis was conducted; No statistical analysis - insufficient study population

ADVERSE EVENTS:
Time Frame: Reported Adverse Events (AEs) for the overall study include events starting on or after study start date and on or before study close date.
Description: Safety population included all participants who received investigational product 99mTc MDP Injection derived from neutron-bombardment. Safety assessments: telephone interview at 14 days, chart check at 30 days.
Groups:
- 99mTc MDP Injection:Fission: Oncologic indication for which a bone scan would normally be indicated.
  99mTc MDP Injection:fission: Technetium (99mTc) Medronate Injection USP labeled with 99mTc derived from fission-sourced 99Mo.
Arm/Group | 99mTc MDP Injection:Fission | 99mTc MDP Injection:Neutron-bombardment
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 0/4 | 0/4

LIMITATIONS AND CAVEATS:
Early termination. Despite a relatively comprehensive review of the first four subject's bone imaging scans a cause of an observed altered biodistribution is not apparent. As such study recruitment will be terminated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes